CLINICAL TRIAL: NCT06350045
Title: Renal Puncture Above the Eleventh Rib (High Supracostal Approach) Versus Subcostal Puncture in Percutaneous Nephrolithotomy for Treatment of Renal Stones in Adults: A Prospective Randomized Trial
Brief Title: High Supracostal Versus Subcostal Puncture in Adult PCNL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Gaber, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: supra 11th puncture PCNL
Record Dates: First submitted 2024-03-29; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: closed envelop
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- subcostal puncture PCNL (Experimental): puncturing the subcostal region to reach the kidney
  Interventions: Combination Product: PCNL
- supracostal puncture PCNL (Experimental): puncturing the supra eleventh rib
  Interventions: Combination Product: PCNL

INTERVENTIONS:
Combination Product: PCNL — percutaneous nephrolithotomy

SUMMARY:
as the supra eleventh puncture PCNL is not well investigated in the literature we will conduct that randomised trial in comparison to the subcostal one

DETAILED DESCRIPTION:
The use of percutaneous nephrolithotomy (PCNL) was first reported by Fernström and Johansson in 1976. Percutaneous nephrolithotomy (PCNL) is the accepted treatment for staghorn stones, large renal stones, and some upper ureteric stones. Achieving suitable access to the appropriate calyx is one of the most important steps during the PCNL procedure. Effective puncture is key for the success of PCNL. An ideal percutaneous nephrolithotomy (PCNL) puncture has been described as one that provides the shortest and straightest access to all calculi, avoids major vessels, bowel and lung, lies along the axis of the calyx and causes minimal parenchymal damage.

Many studies have reported that supracostal access for PCNL is advantageous over infracostal access. By creating a straight path along the kidney's long axis, the upper-pole method guarantees access to the majority of the collecting system and makes it simpler to manipulate the rigid nephroscope and other rigid devices. Therefore, supracostal puncture is perhaps the greatest method for gaining access to the upper pole calyx, where staghorn and big, complicated renal stones are most likely to be located. Although pneumothorax, hydrothorax, and lung damage (1-10%) can result after a supracostal puncture, this injury can now be handled with minimal morbidity thanks to advances in surgical technique and understanding of pleural and diaphragmatic architecture.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients amenable for PCNL with stone burden between 2 cm - 4 cm (guy score 1-2-3)

Exclusion Criteria:

* Ectopic kidney.
* Single middle calyceal stone.
* Skeletal anomalies.
* Bleeding diathesis.
* Active urinary tract infection.
* Patient refusing participation.
* Patients with active pulmonary and pleural disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | within 3 months post operative
  Clavien -Dindo classification.
Stone free rate | within 3 months post operative
  the patient being either completely stone-free or there are residual fragments (less than 4 mm).

SECONDARY OUTCOMES:
duration of Hospital stay. | Postoperativly
  post operative hospital stay
Operative time | intraoperative
  from the puncture until withdrawal of the endoscope at the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: ayman assem, dr, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernstrom I, Johansson B. Percutaneous pyelolithotomy. A new extraction technique. Scand J Urol Nephrol. 1976;10(3):257-9. doi: 10.1080/21681805.1976.11882084. PMID 1006190
- [Background] Galvin DJ, Pearle MS. The contemporary management of renal and ureteric calculi. BJU Int. 2006 Dec;98(6):1283-8. doi: 10.1111/j.1464-410X.2006.06514.x. No abstract available. PMID 17125486
- [Background] He Z, Tang F, Lu Z, He Y, Wei G, Zhong F, Zeng G, Wu W, Yan L, Li Z. Comparison of Supracostal and Infracostal Access For Percutaneous Nephrolithotomy: A Systematic Review and Meta-Analysis. Urol J. 2019 May 5;16(2):107-114. doi: 10.22037/uj.v0i0.4727. PMID 30882159
- [Background] Sampaio FJ. Renal anatomy. Endourologic considerations. Urol Clin North Am. 2000 Nov;27(4):585-607, vii. doi: 10.1016/s0094-0143(05)70109-9. PMID 11098758
- [Background] Sinha M, Krishnappa P, Subudhi SK, Krishnamoorthy V. Supracostal percutaneous nephrolithotomy: A prospective comparative study. Indian J Urol. 2016 Jan-Mar;32(1):45-9. doi: 10.4103/0970-1591.173121. PMID 26941494
- [Background] Mousavi-Bahar SH, Mehrabi S, Moslemi MK. The safety and efficacy of PCNL with supracostal approach in the treatment of renal stones. Int Urol Nephrol. 2011 Dec;43(4):983-7. doi: 10.1007/s11255-011-9916-y. Epub 2011 Mar 11. PMID 21394440